CLINICAL TRIAL: NCT01354691
Title: A 6-Month Prospective, Multi-Center, Double-Blind, Placebo-Controlled, Randomized, Adaptive-Trial-Design Study to Evaluate the Safety and Efficacy of 80mg b.i.d Ladostigil in Patients With Mild to Moderate Probable Alzheimer's Disease
Brief Title: Safety and Efficacy Study of Ladostigil in Mild to Moderate Probable Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avraham Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR100101/CO15570
Record Dates: First submitted 2011-05-01; First posted 2011-05-17 (Estimated); Results first posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2018-07

CONDITIONS: Alzheimer's Disease; Dementia; Memory Loss; Cognitive Impairment
Keywords: Alzheimer's Disease; Dementia; Memory Loss; Cognitive Impairment; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurodegenerative Diseases; Delirium, Dementia, Amnestic, Cognitive Disorders; Mental Disorders; Depression; Anxiety
MeSH Terms: conditions — Alzheimer Disease; Dementia; Memory Disorders; Cognitive Dysfunction; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ladostigil hemitartrate (Experimental): Ladostigil capsules 80 mg
  Interventions: Drug: ladostigil hemitartrate
- Placebo (Placebo Comparator): Placebo capsules
  Interventions: Drug: ladostigil hemitartrate

INTERVENTIONS:
Drug: ladostigil hemitartrate — Final dosage strength of 80mg b.i.d will begin at Day 22 following a 21 day dose escalation phase involving 40mg and 60mg b.i.d dosage strengths. Oral, solid dosage.

SUMMARY:
For many, Alzheimer's disease is the number one medical issue facing our aging society. It is a late onset neurodegenerative disease, frequently under diagnosed, that impairs memory and cognitive performance. There are no known treatments that can either prevent or reverse its progression. Consequently, there still remains a need to evaluate treatments which can better stabilize the symptoms of this disease. These symptoms frequently include decreased functional capacity and negative psychological attributes (e,g, depression, anxiety) in association with the memory and cognition deficits. This current study is being done to assess an investigational compound that has been designed to not only improved the cognitive status of affected patients but to also better manage all symptoms. Hence, the ultimate goal is to provide patients with an improved quality of life by slowing the progression of this neurodegenerative disease

DETAILED DESCRIPTION:
This is a phase II, proof of concept study to evaluate the safety and efficacy of the investigational compound ladostigil versus placebo in mild to moderate Alzheimer's disease patients. The randomized, double-blind, placebo-controlled phase of the trial will be 26 weeks in duration and will involve two cohorts (i.e. one arm receiving ladostigil and one arm receiving placebo). After the initial 26 week period, all participating subjects will receive 26 weeks of treatment with ladostigil (i.e. the open label phase). A total of five territories will be participating in this trial. These include Austria, Croatia, Germany, Serbia and Spain.

ELIGIBILITY:
Inclusion Criteria:

* AD diagnosis according to NINCDS-ADRDA criteria
* Mild to moderate AD according to MMSE 14-24 inclusive
* MRI or CT assessment within 6 months before baseline, corroborating the clinical diagnosis and excluding other potential causes of dementia especially cerebrovascular lesions
* Absence of major depressive disease according to CSDD of less than or equal to 18
* Modified Hachinski Ischemic Scale equal to or below 4
* Education for eight or more years
* Previous decline in cognition for more than six months as documented in patient medical records
* A caregiver available and living in the same household or interacting with the patient daily and available if necessary to assure administration of investigational product
* Patients living at home or nursing home setting without continuous nursing care
* General health status acceptable for participation in a 12-month clinical trial and ability to swallow oral medication
* No history of treatment with rivastigmine
* For patients with either donepezil or galantamine anti-cholinesterase inhibitor treatment prescribed, stopped treatment four weeks prior to screening
* For patients with memantine treatment prescribed, stopped treatment four weeks prior to screening

Exclusion Criteria:

* Other primary degenerative dementias (e.g. dementia with Lewy bodies, fronto-temporal dementia, Huntington's disease, Jacob-Creutzfeldt disease)
* Other neurodegenerative conditions (Parkinson's disease. amyotrophic lateral sclerosis, etc)
* Other central nervous system diseases (severe head trauma, tumors, subdural hematoma, etc)
* A current DSM-IV diagnosis of active major depression, schizophrenia or bipolar disorder
* Seizure disorders
* Other infectious, metabolic or systemic diseases affecting central nervous system (syphilis, present hypothyroidism, present vitamin B12 or folate deficiency, serum electrolytes out of normal range, juvenile onset diabetes mellitus, etc)
* Clinically significant, advanced or unstable disease that may interfere with primary or secondary variable evaluations
* Other unstable, chronic or clinically significant medical conditions involving major organs like kidney, liver, lungs and heart/vasculature
* Hospitalization or change of chronic concomitant medications one month prior to screening or during screening period

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-02; Primary Completion 2012-09 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reinhold Schmidt, MD, Principal Investigator — MEDIZINISCHE UNIVERSITAT GRAZ
Locations (19):
- Austria (4):
  - Medizinische Univeritat Graz, Universitatsklinik fur Neurologie, Auenbruggerplatz 22, Graz
  - Privatordination Horn, HamerlingstraBe 15, Horn
  - Allgemeines Krankenhaus der Stadt Linz, KrankenhausstraBe 9, Linz
  - Privatordination, Lainzerstrasse 20, Wein
- Croatia (6):
  - General Hospital Pula, Negrijeva 6, Pula
  - General Hospital Zabok, Bracak 8, Zabok
  - Clinical Hospital Center Zagreb, Kispaticeva 12, Zagreb
  - Clinical Hospital Dubrava, Avenija Gojka Suska 6, Zagreb
  - Polyclinic Neuron, Salata 12, Zagreb
  - Psychiatric Hospital Vrapce, Bolnicka cesta 32, Zagreb
- Germany (3):
  - Klinische Forschung Hamburg GmbH, Hoheluftaussee 18, Hamburg
  - Klinische Forschung Schwerin GmbH, FriedrichstraBe 1, Schwerin
  - Studienzentrum Nordwest, Lange StraBe 23-25, Westerstede
- Serbia (2):
  - Clinical Centre of Serbia, Dr. Subotica 6, Belgrade
  - Military Medical Academy, Crnotravska 17, Belgrade
- Spain (4):
  - CAE Oroitu Centro Atencion Especializada C/Jata, 9, Algorta
  - Centro Geroinnova Barcelona, Calle Mandoni n 17, Barcelona
  - Fundacio ACE, Institut Catala de Neurosciencies Aplicadas, C/Margues de Sentmenat 35-37, Barcelona
  - Institud d' Assistencia Sanitaria de Girona, Edifici La Republica - C/Dr. Castany, s/n, Salt

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ladostigil Hemitartrate | Placebo
Started | 101 | 99
ITT | 99 | 96
PP | 79 | 75
Completed | 80 | 77
Not Completed | 21 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ladostigil Hemitartrate | Placebo | Total
Number analyzed (Participants) | 101 | 99 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 86 | 84 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.25 (6.73) | 74.28 (6.92) | 74.26 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 60 | 116
  Male | 45 | 39 | 84
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White or Caucasian | 101 | 99 | 200
  Ethnicity: Other | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 28 | 27 | 55
  Serbia | 4 | 2 | 6
  Germany | 9 | 8 | 17
  Croatia | 44 | 45 | 89
  Spain | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: ADAS-Cog: Alzheimer's Disease Assessment Scale-Cognitive Subscale
Description: Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) is a brief neuropsychological assessment used to assess the severity of cognitive symptoms of dementia, The ADAS-Cog consist of 11 questions:
  Word Recall Task Naming Objects and Fingers Following Commands Constructional Praxis Ideational Praxis Orientation Word Recognition Task Remembering Test Directions Spoken Language Comprehension Word-Finding Difficulty
  Item scores are summed.
  Low total scores indicate better cognitive performance. Minimum score 0 is best and maximum is 70 - worst.
  For the purposes of analyses the change from baseline is computed to each administration of the test.
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: score on scale - baseline to endpoint
Arm/Group | Ladostigil Hemitartrate | Placebo
Number analyzed (Participants) | 99 | 96
score on scale - baseline to endpoint | -.27 (5.41) | 0.19 (5.15)
Statistical Analysis 1: Comparison: Ladostigil Hemitartrate vs Placebo; Test type: Superiority; p < 0.67, ANCOVA

2. Secondary Outcome: Neuropsychiatric Inventory (NPI)
Description: The Neuropsychiatric Inventory (NPI) was developed to assess psychopathology in dementia patients. It evaluates 12 neuropsychiatric disturbances common in dementia: delusions, hallucinations, agitation, dysphoria, anxiety, apathy, irritability, euphoria, disinhibition, aberrant motor behavior, night-time behavior disturbances, and appetite and eating abnormalities. The severity and frequency of each neuropsychiatric symptom are rated on the basis of scripted questions administered to the patient's caregiver. Higher the score the more disturbed, lower score is thus better. Minimum score is 0 and maximum is 80.
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: score on scale - baseline to endpoint
Arm/Group | Ladostigil Hemitartrate | Placebo
Number analyzed (Participants) | 99 | 96
score on scale - baseline to endpoint | 2.51 (11.27) | 0.66 (7.90)
Statistical Analysis 1: Comparison: Ladostigil Hemitartrate vs Placebo; Test type: Superiority; p < 0.21, ANCOVA

3. Secondary Outcome: Cornell Scale for Depression in Dementia (CSDD)
Description: The Cornell Scale for Depression in Dementia (CSDD) was developed specifically to assess signs and symptoms of major depression in dementia on the basis of a semi-structured interview of a qualified informant. The CSDD evaluates a broad spectrum of depressive signs and synptoms and includes items from other depression scales. Information is obtained from interview of the caregiver as well as from direct observation and interview of the patient CSDD is a 19 item scale assessing depressive status. Higher score more depression. The scale ranges from 0-no depression to 38 maximum depression.
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: score on scale - baseline to endpoint
Arm/Group | Ladostigil Hemitartrate | Placebo
Number analyzed (Participants) | 93 | 86
score on scale - baseline to endpoint | -0.08 (2.81) | -0.45 (3.28)
Statistical Analysis 1: Comparison: Ladostigil Hemitartrate vs Placebo; Test type: Superiority; p < 0.78, ANCOVA

4. Secondary Outcome: Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL)
Description: The Activities of Daily Living ADCS-ADL is a caregiver-based ADL scale composed of 23 items developed for use in dementia clinical trials. It is designed to assess the patient's performance of both basic and instrumental activities of daily living such as those necessary for personal care, communicating and interacting with other people, maintaining a household, conducting hobbies and interests as well as making judgments and decisions. For each ADL, the caregiver is asked whether the patient attempted the activity during the past four weeks. If the answer is positive, the caregiver is then asked to choose the single most accurate definition of the patient's level of performance. Assessment of functional activity status is a 23 item scale measuring impairment in functioning. The scale total score ranges from 0-profound impairment to 30 normal functioning (no impairments)
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: score on scale - baseline to endpoint
Arm/Group | Ladostigil Hemitartrate | Placebo
Number analyzed (Participants) | 99 | 96
score on scale - baseline to endpoint | -1.88 (9.54) | -1.57 (7.72)
Statistical Analysis 1: Comparison: Ladostigil Hemitartrate vs Placebo; Test type: Superiority; p = 0.83, ANCOVA

5. Secondary Outcome: Mini-Mental State Examination
Description: The MMSE is a frequently used screening instrument for AD drug studies. The instrument provides for evaluation of orientation, memory, attention, concentration, naming, repetition, comprehension, ability to create a sentence and to copy two intersecting polygons. This examination is frequently used by physicians in the original diagnosis of AD, and in its subsequent progression, because it can be easily performed in the routine care of patients. A lower score indicates more cognitive impairment. The highest (best) score is 30. The Mini-Mental State Examination, MMSE, is a 30-point questionnaire measures cognitive impairment to screen for dementia. Items are totaled. The scale ranges from 0-most impairment to 30 (normal) no impairment.
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: change in score - baseline to endpoint
Arm/Group | Ladostigil Hemitartrate | Placebo
Number analyzed (Participants) | 99 | 96
change in score - baseline to endpoint | 0.80 (2.73) | 0.60 (2.59)
Statistical Analysis 1: Comparison: Ladostigil Hemitartrate vs Placebo; Test type: Superiority; p = .77, ANCOVA

ADVERSE EVENTS:
Time Frame: 26 weeks
Description: Enrolled patients Ladostigil 101(100.0%) Placebo 99(100.0%) ITT Population Ladostigil 99(98.02%) Placebo 96(96.97%) PP Population Ladostigil 79(78.22%) Placebo 75(75.76%) Safety Population Ladostigil 100(99.01%) Placebo 98(98.99%)
  one patient discontinued the study in each group before administration of drug that is why the Safety Population is: Ladostigil 100(99.01%) Placebo 98(98.99%)
Arm/Group | Ladostigil Hemitartrate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/100 | 2/98
Serious Adverse Events (participants affected / at risk) | 7/100 | 7/98
Other Adverse Events (participants affected / at risk) | 11/100 | 2/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ladostigil Hemitartrate (N=100) | Placebo (N=98)
ACUTE MYOCARDIAL INFARCT (Cardiac disorders) | 1 (1) | 0 (0)
Brain Stroke (Vascular disorders) | 1 (1) | 0 (0)
Elbow Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Femur fracture subtrochan (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sick Sinus Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sun Stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute Cholecystitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Arthritis left ankle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Obstipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneunomia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
POLYTRAUMATISM (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary Infection (Infections and infestations) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ladostigil Hemitartrate (N=100) | Placebo (N=98)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 2 (3)
Essential hypertension (Cardiac disorders) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No